CLINICAL TRIAL: NCT02974933
Title: Apatinib Mesylate Combined With Pemetrexed in the Treatment of Pretreated Advanced Non-squamous Non-small Cell Lung Cancer ：Single Arm Exploratory Study
Brief Title: Apatinib Mesylate Combined With Pemetrexed in the Treatment of Pretreated Advanced Non-squamous Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuling Ou (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry); Hubei Clinical Research Collaboration Group (Unknown)
Responsible Party: Sponsor-Investigator, Wuling Ou, Deputy Chief Physician, Hubei Cancer Hospital
Organization: Hubei Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HubeiCH
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Nonsmall Cell Lung Cancer
Keywords: apatinib; pemetrexed; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib (Experimental): combined with pemetrexed
  Interventions: Drug: Apatinib combined with pemetrexed

INTERVENTIONS:
Drug: Apatinib combined with pemetrexed — For those pretreated non-squamous non-small cell lung cancer, treat with apatinib 500mg Qd, po.combined with pemetrexed continue until disease progression

SUMMARY:
The purpose of this study is to evaluate the efficacy of apatinib mesylate combined with pemetrexed alone in advanced non-small cell lung cancer patients in the second or second line of treatment of progression-free survival

DETAILED DESCRIPTION:
It is a one-arm study. The progression-free survival will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 years to 70years.
2. Histologically or cytologically confirmed non-squamous non-small cell lung cancer(stage IIIB/IV).
3. Measurable lesions as defined by RECIST criteria.
4. Locally advanced lung cancer cannot treat with surgery, recurrent or metastatic lung cancer
5. ECOG performance status (PS) of 0 to 1.
6. Life expectancy ≥3 months.
7. Informed consent.

Exclusion Criteria:

1. Squamous carcinoma (including adeno-squamous carcinoma), small cell lung cancer.
2. Newly diagnosed Central Nervous System (CNS) metastases that have not yet been definitively treated with surgery and/or radiation.
3. Tumor invade big vessels or close to big vessels (less than 5mm)
4. Obvious cavity or necrosis formed in the tumor
5. Uncontrolled hypertension
6. Myocardial ischemia or infarction more than stage II, cardiac insufficiency.
7. Abnormal coagulation (INR>1.5 or PT>ULN+4, or APTT>1.5 ULN), bleeding tendency or receiving coagulation therapy
8. The active HBV or HCV infection
9. History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix.
10. Hemoptysis, more than 2.5ml daily
11. Thrombosis in 12 months, including pulmonary thrombosis, stoke, or deep venous thrombosis.
12. Unhealed bone fracture or wound for long time
13. Received big surgery, had bone fracture or ulcer in 4 weeks.
14. Urine protein≥++, or urine protein in 24 hours≥1.0g
15. Use of CYP3A4 inhibitor within 7 days or CYP3A4 inducer within 12 days prior to enrollment
16. Have received prior treatment with VEGFR TKI (Bevacizumab is permitted).
17. Pregnant or lactating woman, or woman unwilling to practice contraception during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 4 weeks
  evaluation per 28 days

SECONDARY OUTCOMES:
Overall Survival | 4 weeks
  evaluation per 28 days
disease control rate | 4 weeks
  evaluation per 28 days
objective response rate | 4 weeks
  evaluation per 28 days
Adverse Event | 4 weeks
  evaluation per 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ou wuling, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No